CLINICAL TRIAL: NCT04058730
Title: A Comparative Interventional Study to Evaluate the Role of LRYGBP, LSG and SMM in Patients of Type II DM and BMI Between 27.5 - 32.5 kg / m²."
Brief Title: Comparative Interventional Study to Evaluate the Role of LRYGBP, LSG & SMM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Max Institute of Minimally Access, Metabolic & Bariatric Surgery (Other)
Responsible Party: Principal Investigator, DR PRADEEP CHOWBEY, Chairman- Max Institute of Minimal Access, Metabolic and Bariatric Surgery, Max Institute of Minimally Access, Metabolic & Bariatric Surgery
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAMBS04
Record Dates: First submitted 2018-08-20; First posted 2019-08-15 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LRYGBP (Experimental): Laparoscopic Roux en Y Gastric by pass surgery will be evaluated for patients of Type II DM with BMI between 27.5-32.5 kg/m2 Laparoscopic RYGB is primarily a restrictive procedure with a small element of malabsorption.
  Glycosylated Haemoglobin will be used as a parameter to assess the status of Type II Diabetes for these patients to evaluate the effect of the intervention at 1 month, 3 months, 12 months and 24 months post discharge.
  Interventions: Procedure: Laparoscopic Roux en Y Gastric by pass surgery
- LSG (Experimental): Laparoscopic Sleeve Gastrectomy surgery will be evaluated for patients of Type II DM with BMI between 27.5-32.5 kg/m2 Laparoscopic Sleeve Gastrectomy is a pure restrictive procedure. Glycosylated Haemoglobin will be used as a parameter to assess the status of Type II Diabetes for these patients to evaluate the effect of the intervention at 1 month, 3 months, 12 months and 24 months post discharge
  Interventions: Procedure: Laparoscopic Sleeve Surgery
- SMM (Experimental): Standard Medical Management will be evaluated for patients of Type II DM with BMI between 27.5-32.5 kg/m2 Standard Medical management will be as per the recommendation of ADA 2010 guidelines.
  Glycosylated Haemoglobin will be used as a parameter to assess the status of Type II Diabetes for these patients 1 month, 3 months, 12 months and 24 months post consult
  Interventions: Other: Standard Medical Management

INTERVENTIONS:
Procedure: Laparoscopic Roux en Y Gastric by pass surgery
  Arms: LRYGBP
Procedure: Laparoscopic Sleeve Surgery
  Arms: LSG
Other: Standard Medical Management
  Arms: SMM

SUMMARY:
A Comparative Interventional Study to Evaluate the Role of Laparoscopic Roux-en-Y Gastric Bypass (LRYGBP), Laparoscopic Sleeve Gastrectomy (LSG) and Standard Medical Management (SMM) in Patients of Type II Diabetes Mellitus (DM) and Body Mass Index ( BMI) Between 27.5 - 32.5 kg / m²."

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the role of Laparoscopic Roux-en-Y Gastric bypass(LRYGBP), Laparoscopic Sleeve Gastrectomy (LSG) and Standard medical management in patients of type II diabetes and BMI between 27.5 - 32.5 kg / m²."

* A. Partial Remission
* B. Complete Remission
* C. No Remission

Secondary Objective is to evaluate the role of LRYGB, LSG and SMM on other metabolic disorder parameters like

* Dyslipidemia
* Hypertension
* Waist Circumference

This is a study comparing the role of LRYGB, LSG and SMM in subjects suffering from Type II diabetes mellitus with BMI between 27.5 - 32.5 kg/m². Diabetic patients shall be enrolled as per the inclusion and exclusion criteria. The study treatment will be LRYGB surgery or LSG or SMM in subjects who qualify the inclusion/ exclusion criteria.

Post discharge the study subjects will be followed up at the following intervals:

1 Month, 3 Months 12 Months and 24 Months respectively At follow up subjects shall have an overall clinical examination, adverse events and complication shall be recorded and blood samples for laboratory investigation shall be collected.

Number of Subjects

Planned: 150 qualified subjects

To be Analyzed: 150 qualified subjects

Statistical Methods:

Study Population Male and female subjects 30-60 years of age with Type II Diabetes and BMI between 27.5 - 32.5 kg/m2, who fulfill all the inclusion criteria and do not meet any exclusion criteria will be enrolled into the Study.

Sample Size In this study 150 eligible subjects will be enrolled. One Fifty subjects enrolled would provide the 95% of confidence interval with 10% absolute precision.

Statistical Analysis In this study first normality of the data will be checked. Normally distributed data will be analysed by paired t-test. For non- parametric data Wilcox-on signed rank sum test will be used.

As same Subject will be examined at different time points (more than two time points) the ANOVA of Repeated measures will be used. All tests will be two-tailed and the significance level will be 0.05

ELIGIBILITY:
Inclusion Criteria:

* Age 30 to 60 years at the time of enrollment.
* Type II DM present according to standard diagnostic criteria (ADA 2010) for at least 6 months.
* Body mass Index (BMI) between 27.5 - 32.5 kg / m².
* Waist circumference>90 cm if male; >80cm if female.
* Demonstrated to have inadequate control of diabetes defined as HbA1c >8.0mg/dl
* Patients who have given written informed consent.
* Ability to complete the run in for dietary intake and exercise
* Willingness and ability to comply with the follow up protocol, including returns to the clinical center for visits at 1, 3, 12, 24, months post surgery.

Exclusion Criteria:

* TypeII DM of more than 10 years duration.
* Weight loss of more than 9Kgs in preceding six months.
* Currently pregnant or planning to become pregnant.
* Cancer requiring treatment in the past 5 years
* Active HIV or tuberculosis
* CVD event within 6 months prior to enrollment
* Pulmonary embolus in past 6 months
* CVD manifesting any of the following criteria: unstable angina pectoris or angina pectoris at rest; a history of cardiac arrest; complex ventricular arrhythmia at rest or with exercise; uncontrolled atrial fibrillation(heart rate of 100 beats per minute or more); New York Heart Association Class III or IV congestive her failure; acute myocarditis, pericarditis or hypertrophic myocardiopathy; clinically significant aortic stenosis; left bundle block or cardiac pace maker unless approved by cardiologist, cardiac defibrillator; history of aortic aneurysum or at least 7cm in diameter or aortic aneurysum repair; resting heat rate<45 beats per minute or >100 beats per minute; heart transplantation.
* Serum creatinine >1.4mg/dl(women) or 1.5mg/dl(men)
* History of PE or DVT within 6 months
* Abnormal serum free T4 (>1.8) of thryrotropin (TSH >5.5)
* Bilirubin, aspartate amino transferase (AST) or alkaline phosphatase more than thrice the normal.
* Hospitalization for depression in past 6 months.
* Travel plans that inhibits full participation
* History of bariatric surgery, small bowel resection or extensive large bowel resection
* Chronic treatment with systematic corticosteroids
* Current diagnosis of schizophrenia, or other psychotic disorder, bipolar disorder, alcohol abuse or substance abuse.
* Alcoholic or drug addict ( daily consumption of alcohol >60ml in males and >30ml in females)
* Unstable proliferative retinopathy
* Other medical, psychiatric, or behavioral limitations that in the judgments of the investigators may interfere with study participation or the ability to follow the intervention protocol

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Glycosylated Haemoglobin less than 6.5 mg/dl | immediately after the surgery upto 2 years
  The remission of Type II Diabetes Mellitus will be assessed on the basis of the Glycosylated Haemoglobin levels of the patient post surgery.. At 1 month, 3months, 12months, 24 months after discharge

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Max Institute of Minimal Access Metabolic and Bariatric Surgery, New Delhi
  - Max Institute of Minimal Access, Metabolic & Bariatric Surgery, New Delhi

IPD SHARING:
Plan to Share IPD: No